CLINICAL TRIAL: NCT00082186
Title: TRACLEER® (Bosentan) Pulmonary Arterial Hypertension A Multicenter, Open-label, Single-arm Safety Study to Investigate the Effects of Chronic TRACLEER® Treatment on Testicular Function in Male Patients With Pulmonary Arterial Hypertension
Brief Title: The Effect of Tracleer® on Male Fertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Andrea Lauer, PhD, Actelion
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-402
Record Dates: First submitted 2004-04-30; First posted 2004-05-04 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Bosentan

ARMS (1):
- 1 (Experimental): Oral bosentan tablets
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — Oral bosentan tablets 62.5 mg twice daly for 4 weeks, then 125 mg twice daily for 20 weeks.
  Other Names: Tracleer (R)

SUMMARY:
The objective of the study is to evaluate the effects of chronic TRACLEER® treatment on testicular function via semen analysis in male patients with primary pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Male patients age 18-65 years.
* Bosentan-naïve.
* PPH, WHO functional class III/IV, in need of TRACLEER
* Patients pulmonary arterial hypertension (PAH) secondary to congenital heart disease.
* Written informed consent.

Exclusion Criteria:

* Female
* Patients with PAH secondary to connective tissue vascular diseases or HIV.
* Patients who have undergone a vasectomy.
* Patients with an average baseline sperm concentration < 15 x 10[6]/mL, or any sample with a sperm concentration <= 7.5 x 10[6]/mL.
* Patients with an average baseline sperm motility <20% or normal sperm morphology <5%.
* Body weight < 50 kg.
* Hypotension, defined as systolic blood pressure less than 85 mm Hg.
* AST and/or ALT plasma levels greater than 3 times ULN.
* Hypersensitivity to bosentan or any of the components of the formulation.
* Treatment with glyburide, cyclosporine A or tacrolimus at inclusion or planned during the study.
* Treatment with hormone suppressive agents, including androgens, estrogens, anabolic steroids or glucocorticoids within the past 6 months or planned during the study.
* Current treatment less than 3 months prior to inclusion or planned treatment with prostacyclin or prostacyclin analogues (e.g., Flolanâ or Remodulin).
* Patients who received an investigational drug in the month preceding the study start or who are due to be treated with another investigational drug during the study period.
* Known drug or alcohol dependence or any other factors that will interfere with conduct of the study.
* Any illness other than PPH that will reduce life expectancy to less than 6 months.
* Active cancer.
* Prior treatment with an anti-neoplastic agent or ionizing radiation.
* Hot tub/Jacuzzi use.
* Uncontrolled diseases including diabetes, liver or kidney disease.
* Patients receiving spironolactone (aldactone) less than 3 months prior to inclusion or dose >25 mg/day at baseline or anytime during the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-07; Primary Completion 2007-02 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a mean decrease in sperm concentration to 7.5 x 10[6]/mL or below, without a single sperm concentration ≥ 20 x 10[6]/mL, at 3 or 6 months. This proportion is considered of clinical relevance if greater than 30%. | From baseline to end of study.

SECONDARY OUTCOMES:
Semen volume, sperm motility and sperm morphology change | From baseline to 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lauer, Ph.D., Study Director — Actelion Pharmaceuticals US, Inc.; Maurizio Rainisio, Ph.D., Study Director — Actelion; Frederic Bodin, M.D., Study Director — Actelion

REFERENCES:
- See also: Tracleer approval page at Drugs@FDA.gov — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=TRACLEER